CLINICAL TRIAL: NCT04835584
Title: An Open-Label, Multicenter, Phase 1b/2 Study of the Safety and Efficacy of KRT-232 Combined With a Tyrosine Kinase Inhibitor (TKI) in Patients With Relapsed or Refractory Ph+ Chronic Myeloid Leukemia (CML)
Brief Title: KRT-232 and TKI Study in Chronic Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRT-232-117
Record Dates: First submitted 2021-04-05; First posted 2021-04-08 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Chronic Myeloid Leukemia
Keywords: navtemadlin
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; Dasatinib; nilotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1, KRT-232 combined with TKI (Dasatinib or Nilotinib) in patients with CML-CP (Experimental): KRT-232 will be administered orally, once daily (QD) on Days 1-7 in a 28-day cycle. TKI (dasatinib or nilotinib) will be administered orally, per locally prescribed dose and schedule.
  Interventions: Drug: KRT-232; Drug: Dasatinib; Drug: Nilotinib
- Part 2, Arm A (KRT-232 combined with Dasatinib in patients with CML-CP) (Experimental): KRT-232 will be administered orally, once daily (QD) on Days 1-7 in a 28-day cycle. Dasastinib will be administered orally, per locally prescribed dose and schedule.
  Interventions: Drug: KRT-232; Drug: Dasatinib
- Part 2, Arm B (KRT-232 combined with Nilotinib in patients with CML-CP) (Experimental): KRT-232 will be administered orally, once daily (QD) on Days 1-7 in a 28-day cycle. Nilotinib will be administered orally, per locally prescribed dose and schedule.
  Interventions: Drug: KRT-232; Drug: Nilotinib
- Part 2, Arm C (KRT-232 combined with Dasatinib or Nilotinib in patients with CML-AP) (Experimental): KRT-232 will be administered orally, once daily (QD) on Days 1-7 in a 28-day cycle. Dasatinib or Nilotinib will be administered orally, per locally prescribed dose and schedule.
  Interventions: Drug: KRT-232; Drug: Dasatinib; Drug: Nilotinib

INTERVENTIONS:
Drug: KRT-232 — KRT-232 is an experimental MDM2 inhibitor anticancer drug taken by mouth.
Drug: Dasatinib — Dasatinib is a Tyrosine Kinase Inhibitor anticancer drug taken by mouth.
  Other Names: Dasatinib Zentiva
  Arms: Part 1, KRT-232 combined with TKI (Dasatinib or Nilotinib) in patients with CML-CP; Part 2, Arm A (KRT-232 combined with Dasatinib in patients with CML-CP); Part 2, Arm C (KRT-232 combined with Dasatinib or Nilotinib in patients with CML-AP)
Drug: Nilotinib — Nilotinib is an Tyrosine Kinase Inhibitor anticancer drug taken by mouth.
  Other Names: Tasigna
  Arms: Part 1, KRT-232 combined with TKI (Dasatinib or Nilotinib) in patients with CML-CP; Part 2, Arm B (KRT-232 combined with Nilotinib in patients with CML-CP); Part 2, Arm C (KRT-232 combined with Dasatinib or Nilotinib in patients with CML-AP)

SUMMARY:
This study evaluates KRT-232, a novel oral small molecule inhibitor of MDM2, for the treatment of patients with Ph+ Chronic Myeloid Leukemia (CML) who have relapsed or are refractory or intolerant to a Tyrosine Kinase Inhibitor (TKI).

This study is a global, open label Phase 1b/2 to determine the efficacy and safety of KRT-232 in patients with chronic phase CML (CML-CP) and accelerated phase (CML-AP) who have failed TKI treatments.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1b and Phase 2 Arms A and B: Documented TP53wt, Ph+, BCR-ABL+ CML-CP
* Phase 2 Arm C ONLY: Documented TP53wt, Ph+, BCR-ABL+ CML-AP
* Subject is resistant (relapsed or refractory) and/or intolerant to at least 1 prior TKI.
* Adults ≥ 18 years of age.
* ECOG performance status of 0 to 2
* Adequate hematologic, hepatic, and renal functions

Exclusion Criteria:

* Phase 1b and Phase 2 Arms A and B: Documented Ph+, BCR-ABL+ CML-AP
* Documented Ph+, BCR-ABL+ CML-BC
* Known T315I mutation.
* Prior treatment with MDM2 antagonist therapies.
* Intolerance to current TKI therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Maximum tolerated dose (MTD)/maximum administered dose (MAD) of KRT-232 | 28 Days
  DLTs will be used to establish the MTD/MAD of KRT-232 in combination with dasatinib or nilotinib
Part 2, Arm A and B: Major molecular response (MMR) rate | 6 months
  The proportion of subjects who achieved complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR) according to modified ELN criteria
Part 2, Arm C: Major hematological response (MaHR) rate | 6 months
  The proportion of subjects who achieved MaHR according to modified ELN criteria

SECONDARY OUTCOMES:
CCyR rate | 12 months
  The proportion of subjects who achieved CCyR or PCyR according to modified ELN criteria in Arms A and B
MCyR rate | 47 months
  The proportion of subjects who achieved CCyR or PCyR according to modified ELN criteria in Arm C
Duration of response | 47 months
  DOR (Kaplan-Meier estimate) defined as the time from first observation of response to progression/relapse or death, whichever comes first
Rate of complete hematologic response (CHR) | 47 months
  The proportion of subjects who achieve a CHR according to modified ELN criteria in Arms A and B
Progression-free survival (PFS) in each Arm | 47 months
  PFS is defined as the time from the first treatment dose date to progression/relapse or death, whichever comes first
Overall survival (OS) in each Arm | 47 months
  OS is defined as the time from the first treatment dose date to death from any cause

CONTACTS AND LOCATIONS:
Locations (26):
- United States (5):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Texas Oncology- Sammons CC at Baylor, Dallas, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- France (4):
  - Centre Leon Berard, Lyon
  - APHM Hopital de la Timone, Marseille
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospitalier Lyon Sud, Saint-Genis-Laval
- Italy (4):
  - Policlinico di Milano Ospedale Maggiore | Fondazione IRCCS Ca' Granda, Milan, MI
  - Azienda Ospedaliero - Universitaria Mater Domini, Catanzaro
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori, Meldola FC
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Pratia Onkologia Katowice, Katowice, Poland
- Russia (3):
  - National Medical Research Center of Hematology, Moscow
  - Almazov National Medical Research Center, Saint Petersburg
  - Samara State Medical University, Samara
- South Korea (4):
  - Kyungpook National University Hospital, Daegu
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
- Spain (4):
  - Clínica Universidad de Navarra, Madrid, Navarre
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid